CLINICAL TRIAL: NCT05978934
Title: Determining How Indoor Lighting Affects the Brain Health of Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Well Living Lab, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB 22-005400
Record Dates: First submitted 2023-04-27; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Sleep; Physical Activity; Cognitive Function; Social Isolation
MeSH Terms: conditions — Motor Activity; Social Isolation | interventions — Long Interspersed Nucleotide Elements; inulin trinicotinate monomethochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L1 then L2 followed by L3 lighting condition (Active Comparator): Participants will first experience a static lighting condition (L1) then a dynamic lighting condition (L2). After, participants will experience another dynamic lighting condition (L3) with increased morning brightness compared to L2.
  Interventions: Behavioral: Static Lighting Condition (L1); Behavioral: Dynamic Lighting Condition (L2); Behavioral: Dynamic Lighting Condition (L3)
- L2 then L1 followed by L3 lighting condition (Active Comparator): Participants will first experience a dynamic lighting condition (L2) then a static lighting condition (L1). After, participants will experience another dynamic lighting condition (L3) with increased morning brightness compared to L2.
  Interventions: Behavioral: Static Lighting Condition (L1); Behavioral: Dynamic Lighting Condition (L2); Behavioral: Dynamic Lighting Condition (L3)

INTERVENTIONS:
Behavioral: Static Lighting Condition (L1) — This indoor lighting condition keeps a constant brightness and correlated color temperature.
Behavioral: Dynamic Lighting Condition (L2) — This indoor lighting condition has increased brightness and more blue correlated color temperature in the morning hours followed by decreased brightness and less blue correlated color temperature in the afternoon and evening hours.
Behavioral: Dynamic Lighting Condition (L3) — This exploratory indoor lighting condition matches the same pattern as L2 except the brightness in the morning hours is increased.

SUMMARY:
The goal of this randomized, cross-over, single-site trial followed by an exploratory third intervention is to understand how indoor lighting affects different measures of brain health in older adults living in independent living residences. This is a community based study occurring in a local senior living facility. The main question this study aims to answer is:

- How does the quality of ambient indoor lighting an older adult is exposed to affect measures of brain health, such as sleep quality, physical activity, cognitive function, and social engagement?

Participants will be exposed to three different indoor lighting conditions for 4 weeks each while performing the following tasks:

* Wear a smartwatch throughout the study to measure sleep quality and physical activity
* Wear a small, wearable light sensor to measure light exposure during waking hours
* Perform cognitive assessments throughout the study to detect any changes between each of the lighting conditions
* Complete self-report of surveys to assess independence, social engagement, sleep quality, and mood

Results from these tasks will be compared within and between subjects to assess whether the different lighting conditions affect these different measures of brain health.

ELIGIBILITY:
Inclusion Criteria:

1. At least age 60;
2. Able to wear wearable devices throughout the study;
3. Willing to have their lighting in their kitchen and dining areas changed and controlled for the study;
4. Willing to have environmental sensors placed in their residence;
5. Willing to provide contact information about their primary care provider (PCP); and
6. Able and has capacity to provide informed consent (score > 14.5 based on UBACC consent capacity form).

Exclusion Criteria:

1. Is legally blind
2. Previously renovated their living units and no longer have the standard lighting installation offered by the Senior Living Facility;
3. Currently spend or plan to spend most of their day outside of their residence during the study (i.e., would not experience the indoor lighting intervention for the majority of the study);
4. Plan to travel to a different time zone during the study; or
5. Plan to be away from their residence for more than a week during the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time | Change in total sleep time per night over the course of each condition of the 16-week study.
  Total sleep time per night in minutes as measured daily by a wearable device.
Wake After Sleep Onset | Change in wake after sleep onset per night over the course of each condition of the 16-week study.
  Wake after sleep onset per night in minutes as measured daily by a wearable device.
Sleep State Duration | Change in sleep state duration per night over the course of each condition of the 16-week study.
  Sleep state duration per night in minutes as measured daily by a wearable device.

SECONDARY OUTCOMES:
Sleep Quality | Change in self-reported sleep quality over the course of each condition of the 16-week study.
  Self-report measurement of perceived sleep quality made daily via the Groningen Sleep Quality Survey.
Steps Taken | Change in physical activity in steps per day over the course of each condition of the 16-week study.
  Physical activity in steps per day as measured daily by a wearable device.
Physical Activity | Change in physical activity in minutes per day over the course of each condition of the 16-week study.
  Physical activity in minutes per day as measured daily by a wearable device.
Working Memory | Change in working memory performance over the course of each condition of the 16-week study.
  Task performance on a working memory assessment taken twice weekly.
Task Switching | Change in task switching performance over the course of each condition of the 16-week study.
  Task performance on a task switching assessment taken twice weekly.
Response Inhibition | Change in response inhibition performance over the course of each condition of the 16-week study.
  Task performance on a response inhibition assessment taken twice weekly.
Sustained-Attention Reaction Time | Change in sustain-attention reaction time performance over the course of each condition of the 16-week study.
  Task performance on a sustained-attention reaction time assessment taken twice weekly.
Self-Reported Loneliness | Change in self-reported loneliness over the course of each condition of the 16-week study.
  Self-report measurement of loneliness assessed weekly via the UCLA Loneliness Scale.
Self-Reported Depression | Change in self-reported depression over the course of each condition of the 16-week study.
  Self-report measurement of depression assessed weekly via the Positive and Negative Affect Scale.
Self-Reported Mood | Change in self-reported mood over the course of each condition of the 16-week study.
  Self-report measurement of mood assessed weekly via the Depression, Anxiety, and Stress Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- The Waters on Mayowood, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazurek KA, Li L, Klein RJ, Rong S, Mullan AF, Jones DT, St Louis EK, Worrell GA, Chen CY. Investigating the effects of indoor lighting on measures of brain health in older adults: protocol for a cross-over randomized controlled trial. BMC Geriatr. 2024 Oct 11;24(1):816. doi: 10.1186/s12877-023-04594-7. PMID 39394603